# Racial/ethnic differences in micropatch response

PI: Nicole Brogden IRB ID #: 201708721

# **Project Details**

# I. Project Introduction

I.1 Project to be reviewed by:

IRB-01

I.2 Project Title:

Evaluating racial and ethnic differences in micropore closure rates after micropatch application

I.3 Short Title (optional):

Racial/ethnic differences in micropatch response

- 1.4 Provide a short summary of the purpose and procedures of the study proposed in this IRB application.
  - DO NOT include information on studies not proposed in this application.
  - Use LAY terminology only. This must be easily understandable by IRB community members and nonscientists.
  - DO NOT cut and paste technical abstracts from funding applications that may not be understood by a general audience.

The objective of this study is to define the rate of skin barrier recovery following micropatch treatment (also referred to as a microneedle) in subjects of differing racial/ethnic backgrounds. Subjects will be healthy individuals between the ages of 18 - 50 years. Subjects will be divided into groups based on self-identified racial background and BMI. Following enrollment and consent, 9 sites will be identified on the upper arm. Baseline measurements of hydration, electrical impedance, and water loss will be measured at all sites using noninvasive flat probes. Three sites will be treated with a micropatch containing an array of microneedles (800 micrometers in length), followed by a repeated measurement of water loss and impedance; the sites will then be covered with occlusive material secured with medical tape. Three sites will be covered with occlusive material but will not be treated with a micropatch. The remaining three sites will be untreated and uncovered throughout the study and will serve as measurement control sites. The subjects will return at 24, 48, 72, and 96 hours. At each visit the occlusive coverings will be removed and all measurements will be repeated (excluding the water loss measurements). Fresh occlusive material will be applied after measurements are made.

1.5 Specify your research question(s), study aims or hypotheses (do not indicate "see protocol")

The research question we are seeking to answer is whether there are differences in the time it takes for the skin to completely repair after micropatch application in subjects of different race and ethnicities. We hypothesize that the skin of non-Caucasian individuals will restore barrier function more quickly than in Caucasians.

I.6 Background and significance and/or Preliminary studies related to this project. (do not indicate "see protocol")

Transdermal drug delivery (by way of patches that adhere to the skin and deliver drug in a time-dependent fashion) allows for systemic drug delivery through the skin, while avoiding many of the side effects and challenges associated with oral or intravenous drug delivery. One significant challenge limiting the number of drug compounds that can be transdermally delivered is the hydrophobic nature of the skin, which provides a highly efficient barrier against the absorption of drug molecules. Microneedles are a minimally invasive means of assisting the transport of drug molecules across the skin by creating micron-sized channels (also called micropores) in the skin, thereby increasing its permeability. Many studies have demonstrated that microneedle treatment is relatively painless and well-tolerated by most patients.

Following microneedle treatment, the skin must heal the micropores in order to restore barrier function. In young healthy individuals this process takes approximately 48-72 hours when the skin is covered by an occlusive patch. The timeframe for micropore closure is longer in elderly individuals (>65 years of age), taking several days longer to restore the skin barrier. As evidenced by the differences in micropore closure rate observed with advancing age, biological variation can have a significant effect on the skin's healing properties. There are almost no data available regarding how race and ethnicity affect skin response to microneedle insertion. It is crucial to better understand how the rates of micropore closure vary in different racial/ethnic populations because the potential for variability in drug delivery is high if the recovery timeframes are poorly understood.

A number of drug exposure and response factors can be significantly altered in racial subpopulations; these can include pharmacokinetic dose-proportionality, therapeutic index, bioavailability, steepness of the relationship between dose and response, and genetic polymorphisms in metabolism pathways. Whether or not these differences have an effect when a drug is administered via the skin, specifically with microneedles, is unknown. The most obvious skin difference between individuals of varying race is pigmentation. A number of other significant skin differences exist that cannot be visually observed, including epidermal thickness and reactivity. Mean electrical resistance is significantly higher in Black vs. Caucasian individuals, suggesting that the stratum corneum (outer epidermal layer) is thicker or more cohesive, or both. Decreased transdermal penetration of pharmaceuticals has been observed in Black persons (relative to Caucasian). The barrier of darkly pigmented skin is generally more resistant and recovers more quickly to insult than skin of lighter pigmentation. The epidermis is thicker in Korean and Black vs. Caucasian skin. Asian, Caucasian, and Black individuals also have dissimilar levels of skin reactivity. Additional variables that differ between skin of diverse race/ethnicity include transepidermal water loss, hydration, and sebum content. All of these factors could cause clinically relevant differences in micropore healing and drug exposure.

In this study we will measure hydration to characterize the epidermal properties of individuals of different self-identified races. Measurements of water loss and movement of electrical current (impedance measurements) will be used to evaluate the rate of micropore closure. The skin serves as the primary barrier to loss of water from the body, and disruptions of skin barrier function (as seen with microneedle insertion) result in a significant increase in water loss. The skin also serves as a barrier to the movement of electrical current, and a breach of the skin barrier leads to significant decreases in the impedance measurements. Therefore, both of these serve as surrogate markers of barrier function and can be measured noninvasively.

I.7 Literature cited / references (if attaching a grant or protocol enter N/A).

# II. Research Team

II.1 Principal Investigator

Name E-mail College
Nicole Brogden nicole-brogden@uiowa.edu College of Pharmacy

II.2 Team Members
UI Team Members

| Name | E-mail | College | Contact | Key<br>Prsn | UI<br>COI | VAMC<br>COI | Consent Process<br>Involvement | Deactivated |
|---|---|---|---|---|---|---|---|---|
| Nicole Brogden, PharmD, PHD | nicole-<br>brogden@uiowa.edu | College of<br>Pharmacy | Yes | Yes | No | | No | No |
| Jamie Carr, BA | jamie-carr@uiowa.edu | Inst Clinical &<br>Translational | Yes | Yes | No | | Yes | No |
| Nkanyezi Ferguson, MD, MD | nkanyezi-<br>ferguson@uiowa.edu | Carver College of<br>Medicine | No | Yes | No | | Yes | No |
| Abayomi Tolulope Ogunjimi, PHD | abayomi-<br>ogunjimi@uiowa.edu | Graduate College | No | Yes | No | | Yes | Yes |
| Patrick Ten Eyck, MS | patrick-<br>teneyck@uiowa.edu | Inst Clinical &<br>Translational | No | No | No | | No | No |

## Non-UI Team Members

Name Institution Location FWA Role DHHS Contact Key Prsn UI COI VAMC COI Consent Process Involvement Email

Nothing found to display.

II.3 The Principal Investigator of this study is:

Faculty

II.6 Identify the key personnel. The system will automatically designate the PI and all faculty members on the project as "key personnel." For information about other team members who should be designated as "key personnel" please click on the help information.

Name Is Key Personnel

Nicole Brogden, PharmD, PHD Yes

Jamie Carr, BA Yes

Nkanyezi Ferguson, MD, MD Yes

Abayomi Tolulope Ogunjimi, PHD Yes

Patrick Ten Eyck, MS No

II.5 Select research team member who is the primary contact for study participants.

Jamie Carr

# III. Funding/Other Support

III.1 Funding Sources

Type Source Grant Title The effects of pharmacologic and physiologic and physiologic and physiologic of microneedle drug delivery

Departmental / PI Discretionary

\* new source name

III.2 What type of funding agreement would be completed?

Federal/State/Local Agency/Non-Profit Funded/Other

III.3 Does any member of the research team have a financial conflict of interest related to this project according to the <u>Conflict of Interest in Research</u> policy? If yes, please indicate which members below.

| Name | Has Conflict of Interest |
|--------------------------------|--------------------------|
| Nicole Brogden, PharmD, PHD | No |
| Jamie Carr, BA | No |
| Nkanyezi Ferguson, MD, MD | No |
| Abayomi Tolulope Ogunjimi, PHD | No |
| Patrick Ten Eyck, MS | No |

III.5 What is the current status of this funding source?

Source

**Status Other Status Description** 

US Department of Health & Human Services, National Institutes of Health Awarded

# IV. Project Type

IV.1 Do you want the IRB to give this project

Regular (expedited or full board) review

IV.2 Enter the date you will be ready to begin screening subjects/collecting data for this project. (If you do not have a specified date, add

"upon IRB approval")
Upon IRB approval

IV.3 Are you requesting a <u>waiver of informed consent/authorization</u> (subjects will not be given any oral or written information about the

study)?

No

# V. Other Committee Review

V.1 Does this project involve any substance ingested, injected, or applied to the body?

· Do not answer yes, if the involvement includes a device, wire, or instrument

No

V.2 Are any contrast agents used for any purpose in this study?

No

V.9 Will any subject be asked to undergo a diagnostic radiation procedure (including radiographic, nuclear medicine, DEXA)?

No

V.14 Will any subject be asked to undergo a radiation therapy procedure (including external beam therapy, brachytherapy, or nuclear medicine

therapy)?

No

V.20 Does this project involve the deliberate transfer of recombinant or synthetic nucleic acid molecules, or DNA or RNA derived from recombinant

or synthetic nucleic acid molecules, into one or more human research participant?

No

Will any portion of this project be conducted in the CRU, or does it use any CRU resources?

Yes

V.21

V.22 Will this project use:

- any resource/patients of the Holden Comprehensive Cancer Center
- involve treatment, detection, supportive care, or prevention of cancer

No

V.25.a Will the study involve <u>any</u> of the following activity at UI Health Care, even if subjects or their insurance will not be billed for the item or service, and regardless of the study funding source (including studies with departmental or no funding)?

- Procedures, tests, examinations, hospitalizations, use of Pathology services, use of clinic facilities or clinical equipment, or any patient
  care services, including services conducted in the Clinical Research Unit; or
- Physician services or services provided by non-physicians who are credentialed to bill (ARNPs, Physician Assistants, etc.)

Yes

V.25.b Will there be any procedures or services that may happen as part of a subject's regular medical care and as part of the study?

No

V.25.c Will any study equipment or devices be supplied by a study sponsor?

No

V.25.e Is there or will there be an internal budget for this study?

Yes

V.25.f Is there or will there be an external budget for this study?

Yes

V.26 The study involves Department of Nursing Services and Patient Care nursing, nursing resources or evaluates nursing practices at UI

Health Čare.

No

# VI. Subjects

VI.1 How many adult subjects do you expect to consent or enroll for this project?

VI.2 What is the age of the youngest adult subject?

VI.3 What is the age of the oldest adult subject?

VI.4 What is the percentage of adult male subjects?

VI.5 What is the percentage of adult female subjects?

VI.6 How many minor subjects do you expect to consent or enroll for this project?

#### VI.13 Describe EACH of your subject populations

- Include description of any control group(s)
- Specify the Inclusion/Exclusion criteria for EACH group

Approximately 180 subjects aged 18 - 50 will be consented for the study. Target enrollment is 160 subjects, and we anticipate that there will be subjects who will sign consent but not complete the study.

Inclusion criteria: Subjects will be healthy men and women between 18 - 50 years of age who identify as African American or Black, Asian, Hispanic or Latino, American Indian/Alaska Native, Native Hawaiian/Other Pacific Islander, Caucasian/White, bi-/multiracial.

Exclusion criteria: Unable to give consent; severe general allergies requiring chronic treatment with steroids or antihistamines; previous adverse reaction to microneedle insertion; known allergy or adverse reaction to medical tape/adhesive or aloe vera; any inflammatory diseases of the skin; psoriasis, atopic dermatitis, and blistering skin disorders; diseases associated with altered immune function (including but not limited to: rheumatoid arthritis, diabetes, lupus, HIV/AIDS); any subjects taking medication that impairs the immune system (including but not limited to corticosteroids, TNF inhibitors, monoclonal antibodies, chemotherapy agents); any current malignancy or history of malignancy present at the treatment site; eczema or scaling present at the treatment site; any current inflammation or irritation present at the treatment site (including but not limited to: rash, inflammation, erythema, edema, blisters). Uncontrolled mental illness that would, in the opinion of the physician, affect the subject's ability to understand or reliably participate in the study will also be excluded.

Subjects taking medications in the following therapeutic classes will be excluded: HMGCoA reductase inhibitors ("statins"), oral or topical steroids, oral antibiotics, topical antibiotics at the local treatment site, topical antihistamines at the local treatment site, beta-blockers, and systemic or topical NSAIDS/analgesics. A subject who has recently used oral or topical steroids, antibiotics, antihistamines, or analgesics may be enrolled if more than 5 elimination half-lives of the drug have passed since the last dose (this is a typical parameter in pharmacokinetics, when it is assumed that 99% of drug in the systemic circulation is eliminated after 5 half-lives). The estimated elimination half-life for any specific drug will be obtained from standard pharmacy references such as Micromedex or other comparable references.

Any subjects that are pregnant/nursing will be excluded from participation. Subjects will also be excluded for any condition that would, in the opinion of the PI or physician, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

VI.14 Provide an estimate of the total number of subjects that would be eligible for inclusion in each of your study populations (include your control population if applicable)

It is somewhat difficult to know the total number of subjects that would be eligible for the study because we are recruiting generally healthy individuals (of which there will be a large number in the local community). However, it is reasonable to estimate that perhaps several hundred to a few thousand subjects in this local area may be eligible.

VI.15 Describe how you will have access to each of your study populations in sufficient number to meet your recruitment goals.

> This is a relatively small study with low numbers of subjects per group, so we do not anticipate significant challenges with recruitment. We have previously used mass emails and the Noon News to advertise for our studies and have had excellent results. We will post an advertisement in the UIHC outpatient Dermatology clinic and on the University Cambus system as well.

Do you plan to recruit/enroll non-English speaking people? VI.16

VI.18 Do you propose to enroll any of the following in this study as subjects?

- Employee of the PI or employee of a research team member
- Individual supervised by PI or supervised by member of research team
- Individual subordinate to the PI or subordinate to any member of the research team
- Student or trainee under the direction of the PI or under the direction of a member of the research team

Yes

VI.19 Provide justification for why these subjects must be included in the study.

Individuals working in Dr. Nkanyezi Ferguson's Dermatology clinic (residents, fellows) that meet the inclusion requirements may be enrolled if there are unanticipated challenges with recruitment of our subject population.

VI.20 Will subjects provide any information about their relatives?

| VI.23 | Will anyone (other than the subject) provide you with information about the subject (e.g. proxy interviews)? No |
|---|---|
| VI.26 | Is this project <u>about</u> pregnant women?<br>No |
| VI.27 | Will this project involve fetuses?<br>No |
| VI.28 | Does this project involve adult subjects who may be incompetent or have limited decision-making capacity on initial enrollment into the study? No |
| VI.32 | Does this project involve subjects whose capacity to consent may change over the course of the study? No |
| VI.37 | Does this project involve <u>prisoners as subjects</u> ?<br>No |

# VII.A. Project Description (A)

- VII.A.1
- Where will project procedures take place (check all that apply)?
  Other UI campus site After conclusion of the study documents will be stored in the office of the clinical coordinator in 558 CPB or in B105
  - CRU
  - UIHC Dr. Ferguson's dermatology clinic at UIHC
- VII.A.2 Is this project also being conducted by other researchers at their own sites (e.g. a multi-site collaborative project)?

# VII

VII.B.18

| B. Project De | script | tion (B) |
|---|---|---|
| VII.B.1 | Does t | this project involve any of the following (Check all that apply): |
| | • | <b>Registry</b> – The collection and maintenance of data (not including biologic samples) in which: (1) the individuals in the registry have a common or related condition(s), and/or (2) the individuals in the registry are interested in being contacted for future studies by investigators other than those listed in Section II of this project. (UI Guide) |
| | • | Repository – The collection, storage, and distribution of human biologic samples and/or data materials for research purposes. Repository activities involve three components: (i) the collection of data and/or specimens such as blood, tissue, saliva, etc.; (ii) the storage of data or specimens, and data management function; and (iii) the sharing of data/specimens with recipient investigators other than the original investigators. (paraphrased from OHRP) |
| | • | Expanded Access – A process regulated by the Food and Drug Administration (FDA) that allows manufacturers to provide investigational new drugs to patients with serious diseases or conditions who cannot participate in a clinical trial. Examples of expanded access include non-protocol access to experimental treatments, including protocol exception, single-patient IND, treatment IND, compassionate use, emergency use, continued access to investigational drug, and parallel track (ClinicalTrials.gov & FDA). |
| | • | Clinical (or Treatment) trial – A prospective biomedical or behavioral research study of new treatments, new drug or combinations of drugs, new devices, or new approaches to surgery or radiation therapy. (NIH and ClinicalTrials.gov & FDA) |
| | • 🗸 | Physiology intervention/study — A pharmacologic or measurement study aimed at understanding basic mechanisms of disease and/or of normal human physiology, often without any therapeutic intent (though a clinical trial could include such components, often labeled as "translational" or "basic science" aims.) Measurements in such studies could include, but are not limited to, a blood draw, EKG, EEG, MRI, auditory or sensory testing, checking vital signs, DEXA scans, eye tracking, specimen collection, exercise, fasting, special diets, etc. |
| | • | <b>Behavioral intervention/study</b> – May be used to refer to studies of individual or group behavior. This option does not include drugs, biologics, or devices but could include psychotherapy, lifestyle counseling, behavior modification, etc. |
| | • | <b>Diagnostic trial</b> – Protocol designed to evaluate one or more interventions aimed at identifying a disease or health condition (ClinicalTrials.gov & FDA) |
| | • | Non-clinical – any college/department that would regularly submit to <u>IRB-02</u> |
| | • | Other |
| VII.B.1. | | Provide the NCT (National ClinicalTrials.gov Identifier) number NCT03332628 |
| VII.B.2 | | Does this project involve a <u>drug washout</u> (asking subject to stop taking any drugs s/he is currently taking)?<br>No |
| VII.B.11 | | re a separate, written protocol that will be submitted in addition to this IRB New Project form? (Note: a grant application is not<br>lered to be a protocol) |

Does this project involve testing the safety and/or efficacy of a medical device?

# VII.C. Project Description (C)

VII.C.1 Does this project involve any <u>research on genes or genetic testing/research</u>?

# VII.D. Project Description (D)

# VII.D.1 Check all materials/methods that will be used in recruiting subjects (you will need to attach copies of all materials at the end of the application):

- Use of any information available to the researchers or their colleagues because this person is a patient OR use of any information considered
  to be Protected Health Information (PHI) OR review of patient/clinic records Potential subjects that are seen in the Dermatology clinic at
  UIHC will be pre-screened by members of the research team using the electronic medical record (EMR). This information will be used only
  for determining eligibility and will not be collected or stored.
- Existing Registry/database Subject's that have previously enrolled in other studies related to this application will be sent a letter containing
  information about new study opportunities available. Specifically at this time individuals that have participated in IRB#201806039 will be
  contacted.
- Referral from colleague Dermatologists at UIHC seeing patients who they think qualify for the study may refer subjects to the study
  coordinator for more information.
- · Website Iowa Clinical Research & Trials website
- · Advertisements -
- · Posters -
- E-mail -
- Letter -

# VII.D.2 List the individual data elements you will need to access/use from the patient or clinic records to identify potential subjects for recruitment

Researchers will review the patients' age, BMI, current medications, pregnancy/nursing status, and medical conditions (as listed in section VI.13). This information will not be stored or collected as a part of the research data.

# VII.D.3 Describe why you could not practicably recruit subjects without access to and use of the information described above

The Department of Dermatology at UIHC consists of 13 dermatologists and numerous ARNPs, PAs, and medical students. Up to 100 patients can be seen in one day at the clinic. In addition, the Department of Dermatology also has an Ethnic Skin Care Clinic that offers specialized services for patients of color (defined as skin types IV-VI in the Fitzpatrick Skin Type Classification). Patients of color are minority populations in the state of Iowa, and working with the EMR for patients in these dermatology clinics allows us to review eligibility for patients who might otherwise be difficult to access through general advertising. It is necessary for our research team to be able to determine eligible potential subjects prior to their visit because it would not be feasible for us to speak with every patient that the dermatology clinic sees in one day. By determining eligibility prior to their appointment we will be able to increase the efficacy of our recruitment and maximize the outcomes of our study.

# VII.D.4 Describe why you could not practicably obtain authorization from potential subjects to review their patient or clinic records for recruitment purposes.

Due to the large number of patients seen in the dermatology clinics each day, it is not feasible for us to expect that our research team would be able to meet one on one with each of them every day. None of the information reviewed will be recorded or stored for purposes of the study.

# VII.D.5 Describe plans to protect the identifiers from improper use or disclosure

No subject information reviewed using the EMR will be recorded or stored for purposes of this study. All necessary information will be collected from the subject upon consenting in the study.

# VII.D.6 Describe plans to destroy identifiers at the earliest opportunity consistent with conduct of the research

No subject information or patient identifiers will be recorded for purposes of this study.

# VII.D.7 Does the research team agree that the requested information will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the study, or for other research for which the use or disclosure of the requested information would be permitted by the HIPAA Privacy Rule

# VII.D.8 Will a member of the research team discuss the study with the subject in person prior to the subject agreeing to participate? Yes

## VII.D.9 Describe the physical location where the consent process will take place:

The consent process will take place in a private room in the CRU.

# VII.D.10 Will a member of the research team discuss the study with the subject by phone prior to the subject agreeing to participate? Yes

# VII.D.11 Describe:

Individuals who call the study site after viewing one of our many advertisements (mass email, poster in the dermatology clinic or the Cambus, or the noon news) will be provided a brief overview of the purpose and study procedures. If the individual provides permission, they may be asked questions on a pre-screening survey. These questions will help determine if the subject is likely to meet any of the exclusion criteria. If a subject is interested in study participation and passes pre-screening procedures, they may be emailed a copy of the informed consent and invited to attend an informational session at the CRU where staff will present a detailed discussion of the study rationale, procedures, risks, and benefits. Questions will be solicited.

VII.D.12 Who will be involved in the <u>consent process</u> (including review of consent document, answering subjects' questions)?

Name Consent Process Involvement

HawkIRB 10/29/2020

> Name **Consent Process Involvement** Nicole Brogden, PharmD, PHD No Jamie Carr, BA Yes Nkanyezi Ferguson, MD, MD Yes Abayomi Tolulope Ogunjimi, PHD Yes Patrick Ten Eyck, MS No

#### VII.D.15 Check all materials that will be used to obtain/document informed consent:

Consent Document

#### VII.D.16 Are you requesting a waiver of documentation of consent (either no subject signature or no written document)?

Before the subject gives consent to participate are there any screening questions that you need to directly ask the potential subject to determine

eligibility for the study?

VII.D.19

#### List any screening questions you will directly ask the potential subject to determine eligibility. VII.D.20

Are you between 18 - 50 years of age?

How tall are you?

What do you weigh?

What racial group do you self-identify with? (Subject will be provided a list of examples if clarification is required.)

Do you have any general allergies that require daily treatment with steroids or antihistamines?

Have you ever had any kind of microneedle patch applied to your skin? If so, did you experience any adverse reactions to it?

Do you have a known allergy or adverse reaction to medical tape, Band-Aids, adhesive?

Do you have an allergy to aloe vera?

Do you take prescription medications?

Do you have any chronic or ongoing medical conditions (including skin disorders or pregnancy)?

Screening will be streamlined with the use of a redcap survey found at the following link. https://redcap.icts.uiowa.edu/redcap/surveys/? s=4XJ8CYKNCF

# VII.D.21 Will you keep a screening log or other record that would include information on people who do not enroll in the study?

#### VII.D.22 Describe the information being collected and the purpose for keeping this information.

A screening log will be maintained that will document the first and last name of the prospective participant that was screened, date of screening, phone number if provided, email address if provided, and whether it was a screen failure or if the subject will continue on to the consent process. This information will be kept until all study activities have been completed for all participating subjects. We will keep the screening information because it is not uncommon for individuals to respond to the same advertisements more than once (for example, Noon News) and we want to know if a subject has previously contacted us about the study. The log will be destroyed when all subjects have finished the study.

VII.D.23 Will this information be shared with anyone outside the UI research team members?

#### VII.D.25 After the subject agrees to participate (signs consent), are there any screening procedures, tests, or studies that need to be done to determine if the subject is eligible to continue participating?

#### VII.D.26 List and describe screening

After a subject consents to be in the study, baseline demographic data will be collected including age, DOB, sex, height, and weight, race/ethnicity; information regarding current medical conditions and medications will also be collected. Specifically, the subject's approximate duration of each condition/allergy, what treatments the subject has received, and approximate severity of the conditions will be collected, as well as a current medication list. All of this information will be collected directly from the subject and the subject's medical record will not be reviewed/abstracted for research data.

#### VII.D.27 Discuss how much time a potential subject will have to agree to consider participation and whether or not they will be able to discuss the study with family/friends before deciding on participation.

There is no limit on the time a potential subject may take to consider participation. The only restriction on time is that the subject will only be allowed to participate if the study is still enrolling subjects when they provide consent.

#### VII.D.28 How long after the subject agrees to participate do study procedures begin?

Study procedures can begin immediately after obtaining consent.

#### VII.D.29 Provide a description of the enrollment and consent process for adult subjects

- · Describe each study population separately including control population
- · Include when recruitment and consent materials are used
- Use 3rd person active voice "The Principal Investigator will identify subjects. For example, the principal investigator will identify potential subjects, the study coordinator will discuss the study with subjects over the telephone and schedule the first study visit, etc..."
- Describe the steps that will be taken by the research team to minimize the possibility of coercion or undue influence during the consent

This study will be advertised through the University of Iowa campus-wide email system and through the University of Iowa Health Care "Noon News," a daily announcement flier printed for community and faculty members within the UIHC. We will also be using printed fliers to advertise

the study in Dr. Ferguson's Ethnic Skin Care Clinic at UIHC and on the University Cambus System. Subjects will be recruited through the dermatology clinic based upon screening of the EMR as well as by physician referral. Advertisements will also be hung in the University Services Building and various cultural centers on the University campus (African-American Cultural Center, Latino and Native American Cultural Center, and Asian-Pacific American Cultural Center). Advertisements for this study have been created so that specific subject populations may be better reached via targeted advertisements, in order to meet our enrollment goals. The mass mailing advertisement has been written in this way as well. It is possible that the mass email will be distributed to certain listservs of University students/staff/faculty that meet our specific demographic criteria (specifically race and ethnicity); we will be working with ITS, the registrar and HR to build confidential lists of individuals who will receive this email. These lists will only be exchanged directly between ITS, HR, and the registrar. No member of the research team will have access to any information about individuals being emailed in this manner. The 'lowa Clinical Research & Trials website' is used for recruitment purposes. Interested parties complete a survey showing their interest in participating and a member of the research team reaches out to them upon completion.

Individuals who call the study site will be provided a brief overview of the purpose and study procedures. Prospective participants may be prescreened through a telephone survey or a survey link created by researchers using a data collection tool called RedCap. If a subject is interested in study participation and passes pre-screening procedures, they will be invited to sign an informed consent with a study team member (where they will again be provided overview of the study rationale, procedures, risks, and benefits). An informed consent document will be provided to the subject for review prior to any meeting. If the prospective participant cannot receive an informed consent by email, the individual will be invited to review the document with the study coordinator at UIHC, and must be given the option to schedule a separate meeting to sign the document. This ensures that the individual has the chance to review the material in the informed consent on their own time.

Individuals who contact Dr. Ferguson for information about the study will be provided with a brief description of the study. They will also be provided with an informed consent document for them to review on their own time and will be instructed to contact the study coordinator for more information. Individuals identified prior to their appointment in the dermatology clinic will be invited by their physician or a member of the study team to meet with the study team to learn more about the research opportunity. Prior to their appointments individuals that have been screened by members of the study staff will receive a letter in the mail giving them information about the study and notifying them that they may be eligible to participate in the study. The principal investigator of this study is planning to conduct multiple onsite studies involving microneedles; currently a similar study in production is 201806039. Participants from this study will be sent a letter or email with information about this study instructing them to reach out to the study team if they are interested in participation. There will be no follow up to anyone who is sent a letter or email that does not respond.

Screening for this study will be streamlined with the use of a survey created by the research team (link provided in VII.D.20). The link to this survey will be sent to potential subjects via the Noon News, Mass Email, and the Letter to prior subjects. Participants who complete the survey will provide their email address, and the study team will contact them in response to their answers. The information provided by the individual will be used to determine eligibility and will not be kept or stored by the researcher. All information collected for purposes of this study will be collected during an in-person visit with the potential subject.

It is recognized that the consent process must be carried out in an environment where no coercion is applied and where subjects can be adequately informed of the purpose, nature, procedures, risks and hazards of the study. One of the important features of our screening process is the ability for the prospective participant to review the informed consent on his/her own time, outside of the study site. This additionally demonstrates the reliability of the subject if they schedule a follow-up meeting to sign the informed consent.

VII.D.37 Does the study include any form of deception (e.g., providing participants with false information, misleading information, or withholding information about certain study procedures)?

# Examples:

- Procedure includes a cover story that provides a plausible but inaccurate account of the purposes of the research.
- Participants will be provided with false information regarding the particular behaviors of interest in the research.
- Procedures include a confederate pretending to be another participant in the study.
- · Participants will be told that the research includes completion of a particular task, when in fact, that task will not be administered.
- Study is designed to introduce a new procedure (or task) that participants are not initially told about.
- If yes, a waiver of informed consent must be requested under question IV.3.

No

# VII.E. Project Description (E)

VII.E.1 Will subjects be randomized?

No

VII.E.3 Will any questionnaires, surveys, or written assessments be used to obtain data directly from subjects in this study? Yes

VII.E.4 List all questionnaires, surveys, written assessments and ATTACH each one to the application. (NOTE: You are NOT prohibited from attaching copyrighted materials to this application)

There will be a pre-screening questionnaire and a screening questionnaire to collect information from the subjects. File name: Pre-Screening Questionnaire, Screening Questionnaire

A survey will be utilized to help determine an individuals eligibility to participate in the study. This survey can be found at https://redcap.icts.uiowa.edu/redcap/surveys/?s=4XJ8CYKNCF

- VII.E.5 Does this project involve creating any audiotapes, videotapes, or photographs?
- VII.E.6 Provide a detailed description in sequential order of the study procedures following the consent process DO NOT cut and paste from the Consent Document.

Describe study populations separately if they will be participating in different procedures - include CONTROL population if applicable.

DESCRIBE:

• What subjects will be asked to do/what happens in the study (in sequential order)

• The time period over which procedures will occur

- The time commitment for the subject for individual visits/procedures
- Long-term followup and how it occurs

After a subject consents to be in the study, baseline demographic data will be collected for each subject including age, sex, height, weight, and Fitzpatrick skin type (determined by a member of the study team); information regarding current medical conditions will also be collected. Specifically, the subject's approximate duration of each condition, what treatments the subject has received, and approximate severity of the conditions will be collected, as well as a current medication list. All of this information will be collected directly from the subject and the subject's medical record will not be reviewed/abstracted for research data. After completing the questionnaire a member of the research team will determine if the subject is eligible to continue participating in the study. Subjects will be screened out after this process if their answers to screening questions meet the exclusionary criteria. Consent and screening procedures will require approximately 1 hour.

On the first day of study procedures (Day 0), which may occur on the same day as the consenting process, subjects will first be asked to sit quietly in the CRU for 30 minutes before any study procedures are started, in order for their skin to acclimate to the room temperature and humidity. Nine sites will be identified on the upper arm and marked with a pen. At all marked sites baseline measurements of hydration, colorimetry, transepidermal water loss, and impedance will be measured at each site, using noninvasive flat probes (described below). The probes are attached to a computer that calculates measurement units. Three sites will receive the micropatch treatment (described below), and after treatment the transepidermal water loss and impedance measurements are repeated and the sites will be covered by blank occlusive material secured to the skin with medical tape. Three of the sites will receive no micropatch treatment but will be covered with occlusive material. Three of the sites will serve as controls and will receive no treatment and they will remain uncovered. Study procedures on this first day (Day 0) will require approximately 2 - 3 hours. Hair may be clipped (but not shaved) at the identified sites prior to start of the study procedures, if necessary.

The following procedure will be used to apply the micropatch for each subject:

The micropatch will be placed perpendicularly to the skin surface and the microneedles will be inserted by the application of gentle force to the back of the array (the study team member will apply this gentle pressure with their thumb or use of a hand-held applicator). The pressure will be applied for approximately 10 seconds and then the patch will be removed. The patch will be rotated 45 degrees and the same process will be repeated, in order to create a total of 100 non-overlapping pores. The micropatch treatment will only occur on the first study day.

The following procedure will be used to make the baseline and all following measurements of the 9 identified sites:

Several quick measurements will be made at each site, using noninvasive probes.

- a. Transepidermal water loss (TEWL) will be measured at each site by placing a small probe on the surface of the skin for approximately 1 3 minutes at each site. This measurement will not be repeated after Day 0 procedures.
- b. The hydration level of the skin will be measured at each site by placing a corneometer probe lightly on the skin; each measurement takes less than 1 minute at each site.
- c. The redness and color of the skin will be measured at each site by placing a colorimetry probe on skin for less than 1 minute at each site.
- d. Impedance will be measured using an impedance meter with a series of electrodes. This process takes approximately 2 minutes at each site.

Subjects will be asked to return to the CRU at 24 hour intervals for 4 days (24, 48, 72, and 96 hours) after microneedle insertion. At each of these return visits the baseline measurements will be repeated (excluding TEWL measurements). Occlusive coverings will be removed before measurements are taken, and fresh material will be applied afterwards. Each visit will last approximately 1 1/2 - 2 hours.

Within 2 to 3 days following completion of the study, one of the study team members will follow up with the subject via phone or email to determine if the subject is having any redness or skin irritation at the site of any of the treatments. There is no long-term follow up necessary. The overall time commitment for the subjects is approximately 11 - 14 hours with 5 study days (6 if consent and Day 0 procedures do not occur on same day) over 1 week.

# VII.E.7 Will you attempt to recontact subjects who are lost to follow-up?

No - those lost to followup will not be recontacted

## VII.E.9 Will subjects be provided any compensation for participating in this study?

Yes

VII.E.10 Cash

No

VII.E.11 Gift Card

No

VII.E.12 Check

Yes

VII.E.13 Who will be providing the research compensation check to the subject?

Accounting Services directly via the e-Voucher system

VII.E.16 Other

No

# VII.E.19 Describe the compensation plan including

- · Compensation amount and type per visit
- Total compensation
- Pro-rating for early withdrawal from study

Subjects will receive the following compensation:

Day 1-\$50

Day 2-\$25

Day 3-\$25

Day 4-\$25

Day 5-\$25

Total compensation- \$150

Compensation will be prorated for any subject who does not complete all days of the study. Subjects will only be paid for the study days they complete. Subjects will be paid in one check.

# VIII. Risks

VIII.1 What are the risks to subjects including

- emotional or psychological
- financial
- legal or social
- physical?

In general, microneedle treatments are well tolerated. However, the skin could become irritated from the microneedle insertion or from the adhesives (either on the micropatches used to apply the microneedles and make measurements, or the medical tape used to hold the occlusive material in place). There may be mild discomfort, itching, redness, bruising, or hyper-/hypopigmentation at the treatment sites or where adhesives were in contact with the skin. Loss of confidentiality is also a risk.

# VIII.2 What have you done to minimize the risks?

- If applicable to this study ALSO include:
  - How you (members of your research team at Iowa) will monitor the safety of individual subjects.
  - Include a description of the availability of medical or psychological resources that subjects might require as a consequence of
    participating in this research and how referral will occur if necessary (e.g. availability of emergency medical care, psychological
    counseling, etc.)

During the consent process the subjects will be counseled about the micropatch. The skin will be cleansed thoroughly with alcohol wipes prior to applying the micropatch (cleaning technique similar to that used for insertion of a typical hypodermic needle). They will also be counseled about the possibility of local skin irritation and redness from the adhesive tape. Subjects will be closely observed during the measurements and during treatment with the micropatch; emergency facilities and staff will be available if necessary. Subjects will be instructed to contact a member of the study team if problems arise at any time during their participation in the study (all pertinent contact information will be provided to the subjects). Approximately 2 - 3 days following study completion, a member of the research team will call or email the subject to follow-up and be sure that no irritation or infection has occurred.

The risk of loss of confidentiality will be minimized by keeping all documents in a locked cabinet that is only accessible to members of the research team. All electronic forms of data will be kept on a secure-server supported by the University of Iowa that allows only members of the research team access.

VIII.3 Does this study have a plan to have an individual or committee review combined data from all subjects on a periodic basis (such as summary or aggregate safety and/or efficacy data)?

No

# IX. Benefits

IX.1 What are the direct benefits to the subject (do not include compensation or hypothesized results)?

There are no direct benefits to the subjects.

IX.2 What are the potential benefits to society in terms of knowledge to be gained as a result of this project?

As microneedles have now been commercialized with the introduction of the Fluzone Intradermal vaccine in 2011, it is important to learn how different patient populations respond to microneedle treatment so that this unique drug delivery technique can be developed for other applications. The response of different skin types to microneedle application through a micropatch has not been studied previously, and the knowledge gained from this project will help us to optimize drug delivery systems that are non-invasive and can be used in multiple patient populations.

# X. Privacy & Confidentiality

X.1 What are you doing to protect the <u>privacy</u> interests of the subjects?

No direct patient identifiers will be recorded on data collection material. Instead, subjects will be assigned a subject number on study materials. Only the data necessary to answer the research question will be collected, and all consent processes and study procedures will take place in a private location in the Clinical Research Unit.

X.2 Are you collecting the Social Security Number of any subjects for any purpose?
Yes

X.3 Provide the intended usage of SSN:

• To provide compensation to subjects

# X.4 How will information/data be collected and stored for this study (check all that apply):

- Paper/hard copy records (hard copy surveys, questionnaires, case report forms, pictures, etc.) Hard copies will only be transported by
  members of the research team. Hard copies will be stored in the office of the Clinical Coordinator in C44-P of the ICTS center of UIHC or in
  the office of the Clinical Coordinator in 558 CPB in a locked filing cabinet only accessible to members of the study team. Upon closure of
  the study documents will be stored in the office of the Clinical coordinator in 558 CPB or in B105 and B109 ML.
- Electronic records (computer files, electronic databases, etc.) Electronic results and data (after direct patient identifiers have been removed) will be kept on a password protected shared drive (College of Pharmacy, University of Iowa) that only members of the research team will be able to access.
  - o Name Greg Schwartz
  - o Title IT Director

University Job Classification - Faculty/Staff

- X.5 Do the confidentiality protections indicated above allow only members of the research team to access the data/specimens? Yes
- X.7 Does your study meet the NIH criteria for a <u>Certificate of Confidentiality</u> or will you be applying for Certificate of Confidentiality?

# XI. Data Analysis

## XI.1 Describe the analysis methods you will use, including, if applicable, the variables you will analyze

Descriptive statistics will be used for subject demographics. Each subject will serve as their own control, and paired t-tests will determine differences in TEWL (water loss measurements) from baseline to post-microneedle insertion (this is used to determine if the microneedles adequately breached the skin barrier). For the colorimetry and hydration measurements, each daily measurement will be compared to its baseline at that site using paired t-tests. The percent change in TEWL measurements from baseline to post-microneedle application will be calculated and compared between groups.

The impedance data for this study will be analyzed using similar methods as our previous study. The Z-pores impedance value will be calculated, and Student's t-tests will be used to ensure that micropores where adequately created (demonstrated by a significant decrease in impedance from baseline). Next, Z-pores will be calculated from impedance measurements taken over several hours to days following microneedle treatment (depending on the subject group), and then converted to admittance (admittance is the inverse of impedance). The admittance can demonstrate how "open" the micropores are in a very intuitive manner. If a micropore has a maximum admittance, then the micropore is 100% open. Using this information, we will plot admittance vs. time and calculate a rate constant of micropore admittance (k). The rate constant is then used to calculate the half-life of micropore closure, which thus describes a rate of closure in units of time.

XI.2 Provide the rationale or power analysis to support the number of subjects proposed to complete this study.

There is no data in any population other than Caucasian individuals to guide a formal power analysis. Our calculation of subject number was based on what is feasible for a pilot study to give enough preliminary data for a power analysis later. We plan to enroll subjects into 2 groups, determined by their BMI. Group 1: BMI <29.9; Group 2: BMI >30. Within each group there will be 80 subjects, divided as follows: 10 African American or Black, 10 Hispanic/Latino, 10 Caucasian/White, 20 Asian, and 10 American Indian/Alaskan Native, 10 Native Hawaiian/Other Pacific Islander, 10 bi-/multiracial. The Asian group contains more individuals because this racial/ethnic category encompasses individuals from a very large geographic area (China, Japan, India, Thailand, Korea, etc.) and therefore more subjects may be necessary to see significant trends. We have selected 180 subjects as the number for enrollment to help account for those who will complete the informed consent form but will be screened out afterwards.

## XII. Future Research

XII.1 Do you wish to keep any information about subjects involved with this research project so that members of the current research team may contact them in the future for your own research projects?

Yes

XII.2 Do you wish to keep any information about subjects involved with this research project so that other researchers may contact them for future research?

No

XII.3 List the data or information you will keep:

Name and contact information.

XII.4 Does this project involve storing any data, tissues or specimens for future research?

No